CLINICAL TRIAL: NCT06620471
Title: Assessing the Enhanced Precision: The Value of Impedance in Ultrasound-Guided Nerve Blocks, an Exploratory Prospective Observational Study
Brief Title: Assessing the Enhanced Precision: The Value of Impedance in Ultrasound-Guided Nerve Blocks (Axillary, Interscalene, Popliteal Sciatic), an Exploratory Prospective Observational Study
Status: Recruiting | Type: Observational
Sponsor: Lebanese American University (Other)
Responsible Party: Principal Investigator, Georges Assaf, M.D. Anesthesiologist, Lebanese American University
Other Study IDs: LAUGPNB5372
Record Dates: First submitted 2024-09-21; First posted 2024-10-01 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2024-09

CONDITIONS: Impedance; Axillary Nerve Block; Ultrasound-Guided Nerve Blocks; Interscalene Nerve Block; Popliteal Sciatic Nerve Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

SUMMARY:
Impedance can have an impact on nerve block during loco-regional anesthesia, particularly when using techniques such as nerve stimulation or ultrasound guidance to locate and block specific nerves. Impedance refers to the resistance to electrical current flow within tissue, and it can affect the ability to stimulate nerves or visualize them using ultrasound. The aim of this research is to assess the impedance across different tissue type during an axillary peripheral nerve block (skin, fat, fascia, muscle, nerve). The results of this study would help clinicians performing nerve block to enhance the precision of needle placement, thus increase the success rate of nerve block and reduce adverse events such as intraneural or intravascular injections.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years to 90 years old
* No infection at the injection site
* Patient signed the study consent form
* No contraindications for nerve block
* No allergies to any of the drugs used
* Patient able to communicate effectively

Exclusion Criteria:

* Patients not meeting the inclusion criteria
* Patients with bleeding disorders or undergoing anticoagulation therapy
* Pregnant patients
* Patients with mental incapacity
* Any medical conditions posing severe risks during the procedure

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-14 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Assess the impedance across different type of tissue during axillary nerve block | 3 months
  Measure impedance at different locations, different tissue types and different distances from the nerve (as recorded on the nerve stimulator)

CONTACTS AND LOCATIONS:
Locations (1):
- Lebanese American University Rizk Hospital, Beirut, Beyrouth, Lebanon